CLINICAL TRIAL: NCT02134054
Title: Stavanger University Hospital IBD Study - a Cross Sectional Longitudinal Study on Patients Treated With Biologics
Brief Title: Stavanger IBD Study - Cross Sectional
Acronym: SUSI-CS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Rikshospitalet University Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SUSI-CS_1
Record Dates: First submitted 2014-04-29; First posted 2014-05-08 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Therapeutic drug monitoring; Biological treatment; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard blood sampling Serum sampling - trough/antibodies of biological agent
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biologic: Patients on treatment with biologics (infliximab or adalimumab)

SUMMARY:
In this cross sectional and longitudinal study, patients with inflammatory bowel disease on biological treatment with infliximab or adalimumab will be included.

After inclusion, the dosage of their existing biological therapy will be adjusted following regular trough-level and antibody-level monitoring, according to a treatment algorithm.

Disease activity markers, fatigue and QoL will be assessed during the study. The hypothesis is that therapeutic drug monitoring may improve clinical disease outcome after one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with inflammatory bowel disease on treatment with infliximab or adalimumab of any duration (at least 3 doses)

Exclusion Criteria:

* Inability to consent
* Inability to adhere to treatment protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inflammatory bowel disease established (minimum 3 doses) on treatment with infliximab or adalimumab
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | One Year
  Harvey Bradshaw Index <5 Partial Mayo score <=2

SECONDARY OUTCOMES:
Symptom scoring | One Year
  Harvey Bradshaw Index, Partial Mayo Score. Change after therapeutic drug monitoring.
Inflammatory markers | One year
  C reactive protein, Fecal Calprotectin. Change after therapeutic drug monitoring.
Fatigue scoring | One Year
  Assessed by Fatigue severity scale and Visual analogue scale. Change after therapeutic drug monitoring.

OTHER OUTCOMES:
Healthcare resource utilization | One year
  Registration of
  * Outpatient visits
  * Hospital admissions (days)
  * Sick leave (days)
  * Visits at general practitioner due to IBD activity
  * Endoscopy due to IBD activity

CONTACTS AND LOCATIONS:
Overall Officials: Tore B Grimstad, MD, PhD, Principal Investigator — Stavanger University Hospital, Department of Medicine
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimstad T, Carlsen A, Kvaloy JT, Bolstad N, Warren DJ, Aabakken L, Lundin KEA, Karlsen L, Steinsbo O, Omdal R. Fatigue in Inflammatory Bowel Disease: No Effect of Serum Concentrations of Infliximab, Adalimumab or Anti-Drug Antibodies During Maintenance Therapy. Scand J Immunol. 2025 May;101(5):e70029. doi: 10.1111/sji.70029. PMID 40289444
- [Derived] Carlsen A, Omdal R, Leitao KO, Isaksen K, Hetta AK, Karlsen LN, Aabakken L, Bolstad N, Warren D, Lundin KEA, Grimstad T. Subtherapeutic concentrations of infliximab and adalimumab are associated with increased disease activity in Crohn's disease. Therap Adv Gastroenterol. 2018 Mar 14;11:1756284818759930. doi: 10.1177/1756284818759930. eCollection 2018. PMID 29623105